CLINICAL TRIAL: NCT04855370
Title: Use of Non-invasive Measurement of Cardiac Output and Stroke Volume to Assess Risk and Response to Treatment in Patients With Pulmonary Embolism (PE)
Brief Title: Non-Invasive Measurement of Cardiac Output and Stroke Volume in PE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study device no longer available
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Richard N. Channick, Professor of Medicine, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-002033
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism; Pulmonary Embolus/Emboli; Pulmonary Disease; Pulmonary Embolism and Thrombosis; Pulmonary Embolism Subacute Massive; Pulmonary Embolism Acute Massive
Keywords: Pulmonary Embolism; Non-invasive Hemodynamics; Non-invasive Blood Pressure
MeSH Terms: conditions — Pulmonary Embolism; Embolism; Lung Diseases; Thrombosis

STUDY DESIGN:
Intervention Model Description: This is a single center study to evaluate the use of non-invasive measurement of stroke volume and cardiac output to assess risk and response to treatment in patients with acute pulmonary embolism (PE). We anticipate enrolling a total of 40 subjects at Ronald Reagan UCLA Medical Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients diagnosed with Pulmonary Embolism (Experimental): Patients requiring intensive care unit (ICU) level care with a confirmed diagnosis of pulmonary embolism (PE) by computed tomography (CT) angiogram or endobronchial ultrasound (EBUS) prior to or within 4 hours of initiation of any PE therapy or intervention.
  Interventions: Device: Non-invasive hemodynamic measurements

INTERVENTIONS:
Device: Non-invasive hemodynamic measurements — A patient profile will be set up in the Edwards EV1000 clinical platform by inputting the patient's demographic information. One or two Edwards ClearSight finger cuffs will be placed on the index, middle, and/or ring finger on one hand of the patient. A pressure controller will be secured by a forearm strap where the finger cuffs will be connected to the pressure controller. The pressure controller will be connected to the Edwards EV1000 clinical platform monitor. A heart reference sensor (HRS) will be connected to the pressure controller, a finger cuff, and to the patient at heart level. The Edwards EV1000 clinical platform will calibrate the finger probes, then record measurements for 10-30 seconds every 15 minutes for 12 to 24 hours. If two finger probes are available, measurements will alternate between fingers.
  Other Names: Non-invasive blood pressure (NIBP)

SUMMARY:
Pulmonary embolism impacts over 1 in 1000 adults annually and is the third leading cause of cardiovascular death after heart attack and stroke. The consequence of each PE is widely variable. Physiologically, the morbidity and mortality of PE is ultimately caused by failure of the right ventricle. The acute rise in pulmonary vascular resistance caused by a PE can overwhelm the right ventricle, resulting in a drop in cardiac output and death from failure of the heart to provide vital perfusion. Despite the importance of stroke volume and cardiac output in the current understanding of PE mortality, they are notably absent from risk stratification scores because they historically could only be measured invasively.

Novel non-invasive methods of estimating stroke volume and associated cardiac output have the potential to revolutionize PE risk stratification and care. Non-invasive blood pressure (NIBP) monitors can even measure stroke volume beat to beat, allowing for continuous evaluation of cardiac function. NIBP systems are typically composed of a finger cuff with an inflatable bladder, pressure sensors, and light sensors. An arterial pulse contour is formed using the volume clamp method of blood pressure measurement combined with calibration and brachial pressure reconstruction algorithms. The stroke volume with each heart beat can be estimated as the area under the systolic portion of the blood pressure curve divided by the afterload. NIBP monitors may improve clinical care of PE because they allow for assessment of dynamic cardiac changes in real time. Detection of worsening stroke volume in acute PE could inform providers of impending cardiac collapse, and improvement of stroke volume may function as a positive prognostic factor or marker of therapeutic success. Use of NIBP monitors during acute PE to identify clinically significant changes in cardiac function may advance both PE prognostication and management.

Our clinical study proposes to monitor hemodynamic parameters including stroke volume in patients with acute pulmonary embolism using non-invasive blood pressure monitors. The relationship between hemodynamic parameters and PE outcomes will be assessed, as well as the changes in hemodynamic parameters with PE intervention. To our knowledge, interval monitoring of stroke volume during acute PE with NIBP monitors has never been reported before.

DETAILED DESCRIPTION:
This is a single center study to evaluate the use of non-invasive measurement of stroke volume and cardiac output to assess risk and response to treatment in patients with acute pulmonary embolism (PE). A total of 40 subjects at Ronald Reagan UCLA Medical Center are anticipated to be enrolled.

After informed consent is obtained, the following procedure will be performed:

Patients requiring ICU level care with confirmed diagnosis of PE by CT angiogram or EBUS will be connected to a device that measures hemodynamics non-invasively called the Edwards ClearSight system and Edwards EV1000 clinical platform for 12 to 24 hours. The device is a finger probe worn with a supportive forearm strap. Hemodynamic measurements from the finger cuff will be recorded at intervals. After 12 hours, measurements will be taken if patient comfort and compliance allows.

Patients will be followed through their hospitalization. Standard of care data will be collected from the medical record including vital signs, cardiac monitor recordings, baseline electrocardiogram, central venous pressure (CVP) if available, ventilator settings and measurements, labs (troponin, d-dimer, lactate, pH, complete blood count, basic metabolic panel, B-type natriuretic peptide (BNP) or N-terminal-pro hormone BNP (NT-proBNP), prothrombin time and international normalized ratio (PT/INR), anti-Xa assay, and partial thromboplastin time (PTT)), imaging, interventions performed, therapies administered, discharge outcome and functional status.

As this is a study looking at the feasibility of non-invasive measurement of cardiac output and stroke volume for treating acute pulmonary embolism, study personnel performing the study procedures will not be blinded to the clinical diagnosis and the management of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age.
* The patient must understand and sign informed consent form (ICF).
* Patients requiring intensive care unit (ICU) level care with a confirmed diagnosis of pulmonary embolism (PE) by computed tomography (CT) angiogram or endobronchial ultrasound (EBUS) prior to or within 4 hours of initiation of any PE therapy or intervention.
* If a patient already has non-invasive hemodynamic monitoring by the Edwards system or by other systems, such as the Cheetah NICOM system, as part of their standard of care, this patient can still be enrolled. If the patient is already being followed by another system such as NICOM, the Edwards system would be added to it as long as the patient consents.

Exclusion Criteria:

* BMI < 20 or BMI > 35.
* Height less than 120 cm.
* Diagnosis of atrial fibrillation, moderate to severe aortic or mitral valve insufficiency or stenosis, scleroderma, or end-stage renal disease.
* Patients on extracorporeal membrane oxygenation (ECMO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
stroke volume (SV) | 12-24 hours
  Stroke Volume (SV) is the volume of blood in millilitres ejected from the each ventricle due to the contraction of the heart muscle which compresses these ventricles.
stroke volume index (SVI) | 12-24 hours
  Stroke Volume Index (SVI) relates SV to body surface area (BSA), thus relating heart performance to the size of the individual. The unit of measurement is millilitres per square metre (ml/m2).
cardiac output (CO) | 12-24 hours
  Cardiac Output (CO) is the amount of blood the heart pumps from each ventricle per minute. It is usually expressed in litres per minute (L/min).
cardiac index (CI) | 12-24 hours
  Cardiac index (CI) is the cardiac output proportional to the body surface area (BSA). The unit of measurement is litres per minute per square metre (L/min/m2).
systemic vascular resistance (SVR) | 12-24 hours
  Systemic vascular resistance (SVR) refers to the resistance to blood flow offered by all of the systemic vasculature, excluding the pulmonary vasculature.
  The units for SVR are most commonly expressed as pressure (mmHg) divided by cardiac output (mL/min), or mmHg⋅min⋅mL^-1
blood pressure (BP) | 12-24 hours
  The pressure of the blood in the circulatory system, often measured for diagnosis since it is closely related to the force and rate of the heartbeat and the diameter and elasticity of the arterial walls.
  Systolic Blood Pressure in mmHg Diastolic Blood Pressure in mmHg
heart rate (HR) | 12-24 hours
  The number of heartbeats per unit of time, usually per minute.
  Measured in beats per minute (BPM)

CONTACTS AND LOCATIONS:
Overall Officials: Richard N Channick, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kucher N, Rossi E, De Rosa M, Goldhaber SZ. Massive pulmonary embolism. Circulation. 2006 Jan 31;113(4):577-82. doi: 10.1161/CIRCULATIONAHA.105.592592. Epub 2006 Jan 23. PMID 16432055
- [Result] Prosperi-Porta G, Solverson K, Fine N, Humphreys CJ, Ferland A, Weatherald J. Echocardiography-Derived Stroke Volume Index Is Associated With Adverse In-Hospital Outcomes in Intermediate-Risk Acute Pulmonary Embolism: A Retrospective Cohort Study. Chest. 2020 Sep;158(3):1132-1142. doi: 10.1016/j.chest.2020.02.066. Epub 2020 Mar 31. PMID 32243942
- [Result] Weatherald J, Boucly A, Chemla D, Savale L, Peng M, Jevnikar M, Jais X, Taniguchi Y, O'Connell C, Parent F, Sattler C, Herve P, Simonneau G, Montani D, Humbert M, Adir Y, Sitbon O. Prognostic Value of Follow-Up Hemodynamic Variables After Initial Management in Pulmonary Arterial Hypertension. Circulation. 2018 Feb 13;137(7):693-704. doi: 10.1161/CIRCULATIONAHA.117.029254. Epub 2017 Oct 25. PMID 29070502
- [Result] Sangkum L, Liu GL, Yu L, Yan H, Kaye AD, Liu H. Minimally invasive or noninvasive cardiac output measurement: an update. J Anesth. 2016 Jun;30(3):461-80. doi: 10.1007/s00540-016-2154-9. Epub 2016 Mar 9. PMID 26961819
- [Result] Goldhaber SZ, Bounameaux H. Pulmonary embolism and deep vein thrombosis. Lancet. 2012 May 12;379(9828):1835-46. doi: 10.1016/S0140-6736(11)61904-1. Epub 2012 Apr 10. PMID 22494827
- [Result] Jimenez D, de Miguel-Diez J, Guijarro R, Trujillo-Santos J, Otero R, Barba R, Muriel A, Meyer G, Yusen RD, Monreal M; RIETE Investigators. Trends in the Management and Outcomes of Acute Pulmonary Embolism: Analysis From the RIETE Registry. J Am Coll Cardiol. 2016 Jan 19;67(2):162-170. doi: 10.1016/j.jacc.2015.10.060. PMID 26791063
- [Result] Jimenez D, Aujesky D, Moores L, Gomez V, Lobo JL, Uresandi F, Otero R, Monreal M, Muriel A, Yusen RD; RIETE Investigators. Simplification of the pulmonary embolism severity index for prognostication in patients with acute symptomatic pulmonary embolism. Arch Intern Med. 2010 Aug 9;170(15):1383-9. doi: 10.1001/archinternmed.2010.199. PMID 20696966
- [Result] Marti C, John G, Konstantinides S, Combescure C, Sanchez O, Lankeit M, Meyer G, Perrier A. Systemic thrombolytic therapy for acute pulmonary embolism: a systematic review and meta-analysis. Eur Heart J. 2015 Mar 7;36(10):605-14. doi: 10.1093/eurheartj/ehu218. Epub 2014 Jun 10. PMID 24917641
- See also: Edwards ClearSight system — https://www.edwards.com/healthcare-professionals/products-services/hemodynamic-monitoring/clearsight-system